CLINICAL TRIAL: NCT04266418
Title: The Evaluation of Banana Flower Stamens Extract on Prevention of Benign Prostatic Hyperplasia in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201911062RSA
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): consume 1 sachet per day for 2 months
  Interventions: Dietary Supplement: Placebo
- Banana flower stamens extract (Experimental): consume 1 sachet per day for 2 months
  Interventions: Dietary Supplement: Banana flower stamens extract

INTERVENTIONS:
Dietary Supplement: Placebo — consume 1 sachet per day for 2 months
  Arms: Placebo
Dietary Supplement: Banana flower stamens extract — consume 1 sachet per day for 2 months
  Arms: Banana flower stamens extract

SUMMARY:
To assess the evaluation of banana flower stamens extract on prevention of benign prostatic hyperplasia in adults

DETAILED DESCRIPTION:
This is a double-blind and randomized study. Subjects are informed to consume the samples every day for 2 months. The clinical diagnosis item of benign prostatic hyperplasia (BPH) is evaluated by the doctor. The questionnaires are collected at every visit of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 40-80 years old
2. 7 ≤ IPSS score <19
3. The subject did not take α-blocker or anticholinergic agents in the last 8 weeks. The subject did not take 5α-reductase inhibitor or androgen suppression agents in the last 16 weeks (depending on medical history).
4. The subject isn't diagnosed with cancer
5. The subject is able to read and finish the information on the questionnaire.
6. The subject must read and sign the informed consent form after the study has been fully explained.

Exclusion criteria:

1. The subject has a history of epilepsy or convulsions, liver and kidney disease, cancer, endocrine disease, mental illness, alcohol or drug abuse, and other major organic diseases (depending on medical history).
2. The lower urinary tract urination symptoms of the subject are not related to prostatic hypertrophy (depending on medical history).
3. Residual urine volume > 250 mL (depending on medical history)
4. Subjects have had pelvic radiation therapy or pelvic surgery (including prostate or bladder surgery, but those who only have had a prostate slice can participate in the trial).
5. Subjects have taken sexual hormone preparations including LHRH agonists, anti-androgens, feminine, or Penta-reductase inhibitors (Proscar and Avodart) 16 weeks prior to the trial.
6. Subjects have participated in other clinical trials 12 weeks prior to the trial.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) | Change from baseline IPSS at 4 weeks and 8 weeks
  To measure the severity of lower urinary tract symptoms. Each item is scored 0-5, yielding a total between 0-35.
Change in Prostate volume | Change from baseline prostate volume at 8 weeks
  To measure the volume of prostate measured by ultrasound

SECONDARY OUTCOMES:
International index of erectile function (IIEF) | Change from baseline IIEF at 4 weeks and 8 weeks
  To evaluate male sexual function over the past 6 months. Each item is scored 1-5, yielding a total between 5-25.
Post-voiding residual urine | Change from baseline post-voiding residual urine at 8 weeks
  To measure and compare the amount of urine left in the bladder after urination before and after treatment. Post-voiding residual urine measured by catheterization or non-invasively by ultrasonography.
Maximum flow rate | Change from baseline maximum flow rate at 8 weeks
  To determine peak urine flow rate and average urine flow rate (mL/sec).

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-How Huang, Doctor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan